CLINICAL TRIAL: NCT00000645
Title: A Phase I Dose Escalation Study of Synthetic Hypericin in HIV-Infected Patients With Less Than 300 CD4 Lymphocytes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: VIMRx Pharmaceuticals (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 150; 11125 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — hypericin

INTERVENTIONS:
Drug: Hypericin

SUMMARY:
To determine the maximum tolerated dose (MTD) of hypericin, to define the types of toxicities that may be observed, and to determine what doses of the drug are associated with improvements in virological and immunological surrogate markers of HIV infection. To determine the bioavailability of synthetic hypericin given in 2 percent benzyl alcohol solution.

Hypericin is unlike other drugs presently being used to treat AIDS patients. Hypericin shows anti-HIV activity in test tube experiments.

DETAILED DESCRIPTION:
Hypericin is unlike other drugs presently being used to treat AIDS patients. Hypericin shows anti-HIV activity in test tube experiments.

Each group of eight patients receives a given dose of hypericin by intravenous infusion. Doses are given three times per week for 8 weeks. When all eight patients at a dose level have been entered and four of the eight patients have completed 3 weeks of therapy without evidence of dose-limiting toxicity, additional patients may begin to receive drug at the next dose level. Concurrently, six patients wll participate in an oral-dosing bioavailability study. NOTE: The initial study was stopped secondary to an MTD being reached.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis for Pneumocystis carinii pneumonia (required for patients with CD4+ < 200).
* Symptomatic treatment with analgesics, antihistamines, antiemetics, antidiarrheal agents, or other supportive therapy.
* Short courses (< 10 days) with ketoconazole or fluconazole for oral candidiasis or acyclovir for herpes lesions.
* Topical medications such as clotrimazole troches or nystatin suspensions.

Concurrent Treatment:

Allowed:

* Blood transfusions.

Patients must have HIV infection with CD+4 lymphocyte count of < 300 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded.

* Kaposi's sarcoma requiring systemic therapy.

Concurrent Medication:

Excluded:

* Continued use of opiates or drugs known to induce photosensitivity.

Patients with the following are excluded:

* Active or chronic opportunistic infection at time of study entry that required curative or suppressive therapy.
* Significant liver disease, orthostatic hypotension, cardiac disease, seizure disorder, lymphoma, hypotension.

Prior Medication:

Excluded:

* Zidovudine (AZT), dideoxyinosine (ddI), dideoxycytidine (ddC), interferon, other antiretroviral agents or immunomodulating drugs within 1 month prior to study entry. Ribavirin within 3 months of study entry.
* Ganciclovir (DHPG), antimycobacterial drugs, MAO inhibitors, hypertension-inducing, nephrotoxic, or hepatotoxic drugs within 14 days of entry.
* Cytotoxic chemotherapy within 1 month prior to study entry.

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Study Completion 1994-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentine FT, Study Chair
Locations (3):
- United States (3):
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - NY Univ. HIV/AIDS CRS, New York, New York

REFERENCES:
- [Background] Gulick R, Lui H, Anderson R, Kollias N, Hussey S, Crumpacker C. Human hypericism: a photosensitivity reaction to hypericin (St. John's Wort). Int Conf AIDS. 1992 Jul 19-24;8(2):B90 (abstract no PoB 3018)
- [Background] Mcauliffe V, et al. A phase I dose escalation study of synthetic hypericin in HIV infected patients (ACTG 150). Natl Conf Hum Retroviruses Relat Infect (1st). 1993 Dec 12-16:159
- [Background] Gulick RM, McAuliffe V, Holden-Wiltse J, Crumpacker C, Liebes L, Stein DS, Meehan P, Hussey S, Forcht J, Valentine FT. Phase I studies of hypericin, the active compound in St. John's Wort, as an antiretroviral agent in HIV-infected adults. AIDS Clinical Trials Group Protocols 150 and 258. Ann Intern Med. 1999 Mar 16;130(6):510-4. doi: 10.7326/0003-4819-130-6-199903160-00015. PMID 10075619